CLINICAL TRIAL: NCT02329704
Title: Evaluation Study Between Density Gradient and Swimming Down for Semen Processing
Status: Completed | Type: Observational
Sponsor: Ahmad Mustafa Mohamed Metwalley (Other)
Responsible Party: Sponsor-Investigator, Ahmad Mustafa Mohamed Metwalley, IVF unit director, Al Baraka Fertility Hospital
Organization: Al Baraka Fertility Hospital (Other)
Other Study IDs: AlBarakaSD2
Record Dates: First submitted 2014-12-28; First posted 2015-01-01 (Estimated); Last update posted 2015-01-01 (Estimated); Status verified 2014-12

CONDITIONS: Infertility
Keywords: IUI/AIH; Semen preparation; Semen processing; ICSI/IVF; ART; Density Gradient; Swimming down; hyaluronan affinity testing; Sperm vitality testin
MeSH Terms: conditions — Infertility | interventions — Diff Quik; Cell Movement

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Semen samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Density Gradient processing: Semen portion processed using Density Gradient (80/40 %) Spin on 1200 r.p.m./20min Wash on 1200 r.p.m./5min Rewash on 1200 r.p.m./5min
  then evaluation to be done using : Diff-Quik staining for morphology evaluation Motility Evaluation for grade A and B Concentration (mil/ml) 24 H half life 48 H half life HBA Testing Bacterial contamination
  Interventions: Procedure: Diff-Quik staining for morphology evaluation; Procedure: Motility Evaluation for grade A and B; Procedure: Concentration (mil/ml); Procedure: 24 H half life; Procedure: 48 H half life; Procedure: HBA Testing; Biological: Bacterial contamination
- Swimming down Processing: Semen portion processed using swimming down (100 %) 30 min at room temperature processing for swim down Wash on 1200 r.p.m./5min Rewash on 1200 r.p.m./5min
  then evaluation to be done using : Diff-Quik staining for morphology evaluation Motility Evaluation for grade A and B Concentration (mil/ml) 24 H half life 48 H half life HBA Testing Bacterial contamination
  Interventions: Procedure: Diff-Quik staining for morphology evaluation; Procedure: Motility Evaluation for grade A and B; Procedure: Concentration (mil/ml); Procedure: 24 H half life; Procedure: 48 H half life; Procedure: HBA Testing; Biological: Bacterial contamination

INTERVENTIONS:
Procedure: Diff-Quik staining for morphology evaluation — Papanicolaou stain (haematoxylin, orange G6, and EA50) gives a clear difference between basophilic and acidophilic cell constituents and thereby enables a detailed examination of chromatin pattern, which is useful in the evaluation of sperm morphology and assessment of presence of immature spermatozoa. Cytoplasmic staining can vary between red and green dependent on ionic strength, pH, and composition of the cell department and the stain (OG6 and EA50).
  Morphological assessment for processed portions of semen. As separation process has to minimize the morphological abnormal sperm.
  Other Names: Abnormal forms %
Procedure: Motility Evaluation for grade A and B — The better separation method will insure more progressive sperms after processing.
  Grading using A and B scale scored by (WHO 2010) references.
  Other Names: Motility %
Procedure: Concentration (mil/ml) — count of isolated sperms Using Makler chamber for count of sperm for each portion post processing.
  Other Names: Concentration for final output
Procedure: 24 H half life — percentage of active motile to non motile sperms.
  Microscopic examination for each sample after 24 hours incubation, to evaluate the progressively motile sperm and those non progressive or non motile.
  Other Names: Motility after 24 hours incubation at 37 Dc.
Procedure: 48 H half life — percentage of active motile to non motile sperms.
  Microscopic examination for each sample after 48 hours incubation, to evaluate the progressively motile sperm and those non progressive or non motile.
  Other Names: Motility evaluation after 48hours incubation at 37 Dc.
Procedure: HBA Testing — The Hyaluronic Binding Assay (HBA®) is an important diagnostic tool for suspected male infertility in the analysis of semen. In a matter of minutes the HBA® slide provides an answer to the proportion of mature binding spermatozoa in the sample (The HBA® score %).
  By using HBA slide we can count the physiologically active sperms at each sample and calculate percentage of active sperms with reference to post processing count from 3rd investigating arm.
  Other Names: Sperm physioogical activity evaluation HA binding
Biological: Bacterial contamination — Routine bacterial culture using Blood Agar culture plates for 10 micron finally washed samples, to confirm presence of any bacteria contamination caused by carry over during processing.
  Other Names: Bacterial contamination presence of post processinf samples

SUMMARY:
This study evaluates the quality of sperm produced after semen processing using Density Gradient (DG) and swimming down (SD).

DETAILED DESCRIPTION:
Semen processing to be used for different ART procedures is essential step to isolate dead sperms as well as those abnormally structural or morphology. Semen preparation will maintain to remove the seminal fluids and present cells and contamination pus cells or bacterial cells.

Among different protocols, Density Gradient and swim-up are the most common. For poor motility and number sample Density Gradient is indicated. While final evaluation for produced or separated sperm form processing procedures was not evaluated yet.

Preparation for evaluation study to compare output of main used protocol Density Gradient (DG) with other protocol as swimming down using different study criteria can make more clear evaluation for better processing procedures.

The cases arranged for evaluation were semen samples are within WHO 2010 normal values for motility and count to be more than 5 million/ml. All samples to be divided to two portions for processing by the two preparation techniques.

Post preparation evaluation to be done for the two outputs using: Motility monitoring for 48 hours at 37.0 Dc, abnormal forms, hyaluronan affinity testing and contaminating bacterial growth.

In this study we will show drawback effect of physical and time stress interface applied on sperms during processing, and compare the out put results with that results produced from sperm processed without centrifugation interface or more processing time. As the sperm will separate it self by its natural movement and normal behavior.

Evaluation will be on three categories:

1. The final output quality: as net highly progressive sperms and their count number ( sperm morphology, count and motility): as our results showed more phonologically normal sperm retrieved from SD method with higher count and more percentage of progressively motile sperms.
2. The quality of sperm produced: through monitoring sperm vitality testing or sperm motility power among 2 days at 37.0 Ds. Motility will be evaluated after 24 hours and 48 hours. Both readings showed more decrease in sperm motility and vitality with time consuming with portions processed using density gradient. While portions processed using SD showed significant better readings.

   Another functional activity of sperm post processing is using HBA testing slide, as we evaluate the sperm affinity to hyaluronan. This Testing or assay indicate the physiological activity of sperm still maintained. While it showed HBA higher significant results with swimming down group study.
3. Final evaluation, that are used to present the quality of separation: is monitored using the contamination and carry over effect during semen manipulation and processing. Bacterial contamination using routine culture media (Blood agar) to evaluate 5 microns from each portions for presence and absence of any bacterial cells or during processing and manipulation.

ELIGIBILITY:
Inclusion Criteria:

* Semen with motility more than 10 % according WHO 2010 standers
* Semen with sperm count more than 5 mil/ml according WHO 2010 standers

Exclusion Criteria:

* Semen volume less than 1.0 ml
* Semen with liquefaction time more than 60 min

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Cases arranged for study were submitted for routine semen analysis. Patient agreements collected as consent form signed during sample submission.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2007-05; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
HBA | 1 day
  Affinity is measured according to percentage of non motile sperm produced from 10 µL of processed sample.
Abnormal forms | 1 day
  Percentage normally stained sperms after processing

SECONDARY OUTCOMES:
Final concentration | 1 day
  Concentration was fluctuation according to original motility and concentration, DG
24 Hour motility | 1 day
  Motility evaluation after 37.0 Dc incubation
48 Hour motility | 2 days
  Motility evaluation after 37.0 Dc incubation

OTHER OUTCOMES:
Bacterial contamination | 2 days
  bacterial culture for 5 micron of processed samples to insure absence of bacterial cells.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad M Metwalley, Study Director — Adliyah
Locations (2):
- Al Baraka Fertility Hospital, Manama, Adliyah, Bahrain
- Ibn Sina IVF Center- Ibn Sina Hospital, Sohag, Sohag Governorate, Egypt

REFERENCES:
- [Background] Malvezzi H, Sharma R, Agarwal A, Abuzenadah AM, Abu-Elmagd M. Sperm quality after density gradient centrifugation with three commercially available media: a controlled trial. Reprod Biol Endocrinol. 2014 Dec 2;12:121. doi: 10.1186/1477-7827-12-121. PMID 25466430
- See also: Description: Density Gradient procedures description — http://www.springerprotocols.com/Abstract/doi/10.1007/978-1-62703-038-0_19